CLINICAL TRIAL: NCT00444587
Title: A Multicenter Phase II Trial of Trastuzumab (Herceptin) Continuation in Combination With 2nd-line Chemotherapies After Progression on a 1st-line Chemotherapy Combined With Trastuzumab in Patients With HER2 Positive Metastatic Breast Cancer (Treatment Beyond Progression, TBP)
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With 2nd-Line Chemotherapy in Patients With HER2 Positive Metastatic Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19944
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (2):
- Trastuzumab + 2nd Line Chemotherapy (Experimental)
  Interventions: Drug: Second line chemotherapy; Drug: trastuzumab [Herceptin]
- Only Chemotherapy (Active Comparator)
  Interventions: Drug: Second line chemotherapy

INTERVENTIONS:
Drug: Second line chemotherapy — As prescribed
Drug: trastuzumab [Herceptin] — 6mg/kg iv every 3 weeks
  Arms: Trastuzumab + 2nd Line Chemotherapy

SUMMARY:
This 2 arm study will compare the efficacy and safety of continuation or discontinuation of Herceptin treatment in combination with 2nd line chemotherapy, in patients with HER2 positive metastatic breast cancer whose condition has progressed on 1st line chemotherapy plus Herceptin. Patients will be randomized either to continue or discontinue Herceptin treatment (6mg/kg iv infusion every 3 weeks) while receiving second-line chemotherapy of the investigator's choice. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >= 18 years of age;
* metastatic breast cancer;
* HER2 overexpression (IHC 3+ and/or FISH positive);
* disease progression during or after previous 1st line chemotherapy + Herceptin;
* scheduled to receive 2nd line chemotherapy.

Exclusion Criteria:

* concurrent immunotherapy or hormonal therapy;
* anthracyclines as part of previous 1st line chemotherapy or planned 2nd line chemotherapy;
* cardiac toxicity during previous 1st line chemotherapy + Herceptin;
* history of other malignancy within last 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Sofia, Bulgaria
- Tallinn, Estonia
- Hungary (8):
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Nyíregyháza
  - Szeged
  - Székesfehérvár
  - Szombathely
- Israel (8):
  - Haifa
  - Holon
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Safed
  - Tel Aviv
  - Ẕerifin
- Lithuania (2):
  - Kaunas
  - Vilnius
- Skopje, North Macedonia
- Slovakia (2):
  - Bratislava
  - Košice
- Turkey (Türkiye) (2):
  - Adana
  - Ankara

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 114 participants were enrolled in this study conducted from March 2007 to August 2011 at 30 centers in 8 countries.
Pre-assignment Details: Of 114 participants screened, 3 participants were screening failures. The reasons for screening failure were violation of inclusion criteria, refused to take part in the study and bacterial infection. Therefore, 111 participants were randomized to receive study treatment. Two participants were randomized but never started study treatment.
Groups:
- Trastuzumab + 2nd Line Chemotherapy: Eligible participants were administered trastuzumab (Herceptin) 6 milligrams per kilograms (mg/kg) of body weight (except in Israel, where the dose was 2 mg/kg body weight), intravenous (IV) infusion every three weeks until disease progression, unacceptable toxicities, or withdrawal from study, in combination with second line chemotherapy.
- Only Chemotherapy: Eligible participants were administered second line chemotherapy according to the investigator's decision.
Period: Overall Study
Arm/Group | Trastuzumab + 2nd Line Chemotherapy | Only Chemotherapy
Started | 93 | 16
Completed | 10 | 1
Not Completed | 83 | 15
Not completed — Death | 2 | 1
Not completed — Progression of the disease | 73 | 8
Not completed — Refused treatment/did not cooperate | 4 | 1
Not completed — Investigator decision | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Missing | 0 | 5

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who entered the trial and received at least one dose of trial medication.
Groups:
- Trastuzumab + 2nd Line Chemotherapy: Eligible participants were administered trastuzumab 6 mg/kg of body weight (except in Israel, where the dose was 2 mg/kg body weight), IV infusion, every three weeks until disease progression, unacceptable toxicities, or withdrawal from study in combination with second line chemotherapy.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + 2nd Line Chemotherapy | Only Chemotherapy | Total
Number analyzed (Participants) | 93 | 16 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.8) | 56.3 (10.2) | 55.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 16 | 109
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Disease Progression
Description: Time to disease progression (TTP) in days was defined as the time from enrollment to objective disease progression (all categories other than objective disease progression was set to be censored including death before progression). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions. Tumor assessments were performed using computer tomography or magnetic resonance imaging. TTP as assessed by investigator, along with a recalculation done by computer algorithm is presented below. Median time was not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Up to 5 years
Population: The Full-Analysis-Set included all participants who were enrolled and had at least one valid primary efficacy variable on active treatment. n = Numbers of participants included in this analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 73
Days
  By Computer (n = 65) | 171 [136 to 322]
  By Investigator (n = 73) | 171 [136 to 265]

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants with tumor shrinkage of a predefined amount. It is a combination of complete response (CR) and partial response (PR) and was assessed according to the RECIST criteria 1.0. Complete response refers to the disappearance of all target lesions and all non-target non-measurable lesions. Partial Response refers to an at least 30 percent decrease in the sum of longest diameter of target lesions, taking as reference the baseline sum longest diameter. Objective response rate was not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Up to 5 years
Population: The Full-Analysis-Set participants with measurable disease with CR or PR
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Trastuzumab + 2nd Line Chemotherapy: Eligible participants were administered trastuzumab 6 mg/kg of body weight (except in Israel, where the dose was 2 mg/kg body weight), intravenous infusion, every three weeks until progression or withdrawal, in combination with second line chemotherapy.
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 87
Percentage of participants
  By Investigator (n= 87) | 43.7 [33.1 to 54.8]
  By computer (n=87) | 43.7 [33.1 to 54.8]

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) was defined as the percentage of participants taking a benefit from the treatments. CBR includes 1) Complete response (CR): disappearance of all target lesions and all non-target non-measurable lesions 2) Partial response (PR) : >=30% decrease in the sum of the longest diameter of target lesions and 3) Stable disease (SD): non-PR and non-progressive disease. It was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST 1.0) and assessed by CT or MRI by the investigator. CBR was also assessed by computer. Clinical benefit rate was not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Up to 5 years
Population: The Full-Analysis-Set participants with measurable disease with CR, PR and SD. Study design was changed to single arm study because herceptin use after progression herceptin-based therapy become widespread.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 87
Percentage of participants
  By Computer (n = 87) | 75.9 [65.5 to 84.4]
  By Investigator (n = 87) | 72.4 [61.8 to 81.5]

4. Secondary Outcome: Median Time to Treatment Failure
Description: Time to treatment failure is defined as a composite endpoint measuring time (number of days) from enrollment to discontinuation of treatment or change in treatment for any reason, including disease progression, treatment toxicity and death. Median time to treatment failure was not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Up to 5 years
Population: The Full-Analysis-Set included all participants who were enrolled and had at least one valid primary efficacy variable on active treatment. Only those participants who experienced treatment failure were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 80
Days | 154 [131 to 238]

5. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time (number of days) between enrollment and the date of death due to any cause. Overall survival was not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Up to 5 years
Population: The Full-Analysis-Set included all participants who were enrolled and had at least one valid primary efficacy variable on active treatment. Only those participants with data available were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 41
Days | 717 [589 to 1057]

6. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant who is administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Trastuzumab + 2nd Line Chemotherapy | Only Chemotherapy
Number analyzed (Participants) | 93 | 16
Number of participants
  Number of participants with any AE | 84 | 10
  Number of participants with any SAE | 20 | 2

7. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Mean Serum Glutamic Oxaloacetic Transaminase, Serum Glutamic-pyruvic Transaminase and Alkali Phosphatase Levels
Description: Participants in the study were evaluated for the serum glutamic oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT) and alkali phosphatase (ALP) at Visit 1 and final study assessments (Up to 5 years). Serum glutamic oxaloacetic transaminase, Serum glutamic-pyruvic transaminase and Alkali Phosphatase levels were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and Final study Assessments (Up to 5 years)
Population: The Safety Population included all participants who entered the trial and received at least one dose of trial medication. n = the number of participants analyzed at a given time point.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 93
Units per liter
  SGOT, Visit 1, (n = 93) | 31.46 (29.78)
  SGOT, Final study assessments, (n = 62) | 36.16 (34.91)
  SGPT, Visit 1, (n = 93) | 25.86 (20.55)
  SGPT, Final study assessments, (n = 61) | 28.19 (16.92)
  ALP, Visit 1, (n = 93) | 202.30 (149.98)
  ALP, Final study assessments, (n = 62) | 193.49 (148.11)

8. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Mean Total Bilirubin and Serum Creatinine Levels
Description: Participants in the study were evaluated for the total bilirubin and serum creatinine. Total Bilirubin and serum creatinine levels were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and Final study Assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Micromole/liter
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 93
Micromole/liter
  Total bilirubin, Visit 1, (n = 93) | 13.50 (42.74)
  Total bilirubin, Final study assessments(n = 60) | 19.16 (36.77)
  Serum creatinine, Visit 1, (n = 92) | 81.18 (61.75)
  Serum creatinine,Final study assessment (n = 63) | 82.53 (70.86)

9. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Mean Albumin Levels
Description: Participants in the study were evaluated for the albumin at Visit 1 and Final study assessments. Albumin levels were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and Final study assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 84
gram per liter
  Albumin, Visit 1, (n = 84) | 43.99 (3.29)
  Albumin, Final study assessments, (n = 54) | 41.07 (6.96)

10. Secondary Outcome: Biochemistry Safety Laboratory Parameters: Mean Urea, Sodium and Potassium Levels
Description: Participants in the study were evaluated for the biochemical safety laboratory parameters urea, sodium and potassium. Urea, sodium and potassium levels were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and Final study assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Millimole per liter
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 92
Millimole per liter
  Urea, Visit 1, (n = 92) | 6.33 (3.07)
  Urea, Final study assessments, (n = 63) | 6.92 (4.93)
  Sodium, Visit 1, (n = 92) | 140.58 (3.34)
  Sodium, Final study assessments, (n = 61) | 139.16 (3.71)
  Potassium, Visit 1, (n = 91) | 4.40 (0.45)
  Potassium, Final study assessments, (n = 61) | 4.22 (0.40)

11. Secondary Outcome: Hematology Safety Laboratory Parameters: Mean Hemoglobin Levels
Description: Participants in the study were evaluated for the Hemoglobin up to 5 years. Hemoglobin levels were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and final study assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 93
grams per deciliter
  Hemoglobin, Visit 1, (n = 93) | 12.67 (2.03)
  Hemoglobin, Final study assessments, (n = 67) | 11.00 (3.57)

12. Secondary Outcome: Hematology Safety Laboratory Parameters: Mean Total Leukocytes Counts
Description: Participants in the study were evaluated for the total leukocytes up to 5 years. Total leukocytes counts were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and final study assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 leukocytes/L
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 92
10^9 leukocytes/L
  Total Leukocytes, Visit 1, (n = 92) | 8.00 (8.60)
  Total Leukocytes, Final study assessment (n =67) | 7.53 (6.88)

13. Secondary Outcome: Hematology Safety Laboratory Parameters: Percent of Differential for Neutrophils, Basophils, Eosinophils, Lymphocytes and Monocytes Counts
Description: Participants in the study were evaluated for the Neutrophils, Basophils, Eosinophils, Lymphocytes and Monocytes at Visit 1 and final study assessments.
  Neutrophils, Basophils, Eosinophils, Lymphocytes and Monocytes counts were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and final study assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent of differential
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 93
percent of differential
  Neutrophils, Visit 1, (n = 93) | 64.89 (10.66)
  Neutrophils, Final study assessments, (n = 64) | 62.22 (14.80)
  Basophils, Visit 1, (n = 86) | 0.38 (0.33)
  Basophils, Final study assessments, (n = 59) | 1.28 (6.34)
  Eosinophils, Visit 1, (n = 88) | 2.36 (2.15)
  Eosinophils, Final study assessments, (n = 61) | 2.50 (3.56)
  Lymphocytes, Visit 1, (n = 93) | 26.34 (9.37)
  Lymphocytes, Final study assessments, (n = 64) | 26.48 (12.85)
  Monocytes, Visit 1, (n = 89) | 5.92 (2.22)
  Monocytes, Final study assessments, (n = 59) | 7.25 (3.56)

14. Secondary Outcome: Hematology Safety Laboratory Parameter: Mean Platelets Counts
Description: Participants in the study were evaluated for the platelets at Visit 1 and final study assessments. Platelet counts were not assessed for 'Only Chemotherapy' group as randomization of participants was not feasible considering Trastuzumab widespread use in routine clinical practice.
Time Frame: Visit 1 [Screening Period (6 weeks prior to enrollment)] and final study assessments (Up to 5 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Number of cells x 10^9/L
Arm/Group | Trastuzumab + 2nd Line Chemotherapy
Number analyzed (Participants) | 93
Number of cells x 10^9/L
  Platelets, Visit 1, (n = 93) | 263.14 (63.91)
  Platelets, Final study assessments, (n = 67) | 256.64 (78.64)

15. Secondary Outcome: Mean Left Ventricular Ejection Fraction
Description: Left ventricular ejection fraction (LVEF) is a measure of the percent of blood ejected from the ventricle in one heartbeat. It is a measure of cardiac function and was assessed by echocardiogram or multigated angiogram at Visit 0 [Screening period (6 weeks prior to enrollment)] and final study assessments (Up to 5 years).
Time Frame: Visit 0 [Screening period (6 weeks prior to enrollment)] and final study assessments (Up to 5 years).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent of blood pumped from LV chamber]
Groups:
- Only Chemotherapy: Eligible participants received second line chemotherapy according to the investigator's decision.
Arm/Group | Trastuzumab + 2nd Line Chemotherapy | Only Chemotherapy
Number analyzed (Participants) | 92 | 16
percent of blood pumped from LV chamber]
  Visit 0 (n = 92, 16) | 63.3 (6.8) | 62.6 (6.9)
  Final study assessment (n= 53, 5) | 61.2 (7.4) | 68.6 (5.9)

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: The Safety Population included all participants who entered the trial and received at least one dose of trial medication.
Arm/Group | Trastuzumab + 2nd Line Chemotherapy | Only Chemotherapy
Serious Adverse Events (participants affected / at risk) | 20/93 | 2/16
Other Adverse Events (participants affected / at risk) | 81/93 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + 2nd Line Chemotherapy (N=93) | Only Chemotherapy (N=16)
Granulocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 2 | 0
Retinal detachment (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + 2nd Line Chemotherapy (N=93) | Only Chemotherapy (N=16)
Agranulocytosis (Blood and lymphatic system disorders) | 5 | 0
Anemia (Blood and lymphatic system disorders) | 25 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 76 | 3
Neutropenia (Blood and lymphatic system disorders) | 80 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 4 | 0
Cardiac failure (Cardiac disorders) | 6 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 4 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 0
Keratitis (Eye disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 52 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 53 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 21 | 1
Asthenia (General disorders) | 15 | 0
Chest pain (General disorders) | 3 | 0
Chills (General disorders) | 2 | 0
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 30 | 7
Gait disturbance (General disorders) | 4 | 0
Infusion site inflammation (General disorders) | 2 | 0
Infusion site pain (General disorders) | 7 | 0
Local swelling (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 8 | 4
Pain (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 2 | 1
Pyrexia (General disorders) | 11 | 0
Hypersensitivity (Immune system disorders) | 4 | 0
Bronchitis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 2 | 0
Eye infection (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 2 | 0
Ejection fraction decreased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Dizziness (Nervous system disorders) | 13 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 8 | 0
Hypoaesthesia (Nervous system disorders) | 10 | 0
Neuropathy peripheral (Nervous system disorders) | 5 | 3
Paraesthesia (Nervous system disorders) | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Polyneuropathy (Nervous system disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 37 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 19 | 1
Phlebitis (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.